CLINICAL TRIAL: NCT02129517
Title: Oncology Nurse IMPACT: Improving Communication With Patients About Clinical Trials
Brief Title: Web-Based Tailored Educational Program in Improving Nurse Communication With Patients About Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE2Z14; NCI-2014-00829 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE2Z14 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Healthy, no Evidence of Disease
MeSH Terms: interventions — Methods; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (IMPACT Intervention) (Experimental): Oncology nurses watch tailored, web-based informational video clips addressing knowledge, attitudes, subjective norms, and perceived behavioral control (barriers of discussing clinical trials with patients). They also watch role-play video clips to help improve perceived behavioral control and address attitudinal barriers.
  Interventions: Other: IMPACT intervention; Other: survey administration
- Arm II (online educational materials) (Active Comparator): Oncology nurses view online clinical trials educational materials developed based upon NCI clinical trials educational materials for health care providers. The educational materials contain text and tables as presented on the NCI Website.
  Interventions: Other: Online education materials; Other: survey administration

INTERVENTIONS:
Other: IMPACT intervention — Tailored, web-based educational short video clips
  Other Names: intervention, educational; educational intervention
  Arms: Arm I (IMPACT Intervention)
Other: Online education materials — Online NCI-based educational materials
  Other Names: intervention, educational
  Arms: Arm II (online educational materials)
Other: survey administration — Ancillary studies

SUMMARY:
This pilot, randomized clinical trial studies a web-based tailored educational program in improving nurse communication with patients about clinical trial treatment options. A web-based tailored educational program may empower and prepare nurses to discuss clinical trial treatment options with patients and may also increase patient participation in clinical trials.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop and pilot test a theory-driven, web-based, tailored, interactive educational program (Oncology Nurse IMPACT: Improving Communication with Patients about Clinical Trials) for oncology nurses to address barriers to discussing clinical trials with patients.

II. To implement Oncology Nurse IMPACT on a national level and conduct a formal program evaluation.

III. To evaluate the mediators and moderators of education program effect on intentions to discuss clinical trials with patients.

OUTLINE: Participants are assigned to 1 of 2 intervention arms.

ARM I: Oncology nurses watch web-based informational video clips addressing knowledge, attitudes, subjective norms, and perceived behavioral control (barriers of discussing clinical trials with patients). They also watch role-play video clips to help improve perceived behavioral control and address attitudinal barriers.

ARM II: Oncology nurses view online clinical trials educational materials developed based upon National Cancer Institute (NCI) clinical trials educational materials for health care providers. The educational materials contain text and tables as presented on the NCI Website.

After completion of study intervention, participants are followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Currently practicing nurse
* Involved in direct patient care
* Self-identify in one of the following primary practice roles--case managers, clinical nurse specialists, nurse practitioners, managers/coordinators, nurse navigators, patient educators, and staff nurses
* Available email address

Exclusion Criteria:

* Research nurses, nurses without direct patient care, and nurse managers/directors (i.e. not involved in direct patient care)
* Lack of email address

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1262 (Actual)
Dates: Start 2014-11-07 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Change in nurse's intention to discuss clinical trials with patients | Baseline to 3 months post-intervention
  Behavioral intention will be assessed using 4 items (3 with 7 point scales, strongly agree/strongly disagree and 1 which asks for an estimated number of patients). An analysis of covariance (ANCOVA) will be used to compare intention scores, adjusting for the pre-intervention intention score as well as age, ethnicity, education, access to clinical trials, and years spent in nursing as well as other key factors found to be significantly imbalanced between groups.

SECONDARY OUTCOMES:
Change in knowledge, attitudes, normative beliefs, and perceived behavioral control | Baseline to 3 months post-intervention
  Actual behavior will be measured using a 3-item scale asking participants to provide an estimate of how many patients they spoke with about cancer clinical trials in the past three months (3-month follow-up) and over the past week (subset of nurses completing the biweekly ecological momentary assessment surveys). An ANCOVA approach will be used to examine effects of the intervention on knowledge, attitudes, behavioral control and normative beliefs.

OTHER OUTCOMES:
Number of patients enrolled in clinical trials | Up to 3 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Neal Meropol, MD, Principal Investigator — Case Comprehensive Cancer Center; Barbara Daly, PhD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Flocke SA, Nock NL, Fulton S, Margevicius S, Manne S, Meropol NJ, Daly BJ. A National Study of Oncology Nurses Discussing Cancer Clinical Trials With Patients. West J Nurs Res. 2019 Dec;41(12):1747-1760. doi: 10.1177/0193945919829145. Epub 2019 Feb 19. PMID 30782111